CLINICAL TRIAL: NCT06991790
Title: A Prospective, Single-arm, Multicenter Phase II Clinical Study of Sacituzumab Govitecan in Combination With Toripalimab as First-line Treatment for Advanced Triple-negative Breast Cancer and an Exploratory Study of Biomarkers for Predicting Efficacy
Brief Title: Sacituzumab Govitecan + Toripalimab as First - Line Therapy for Advanced Triple - Negative Breast Cancer and Biomarker Exploration
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, songguohong, Chief Physician, Deputy Director of the Department, Medical Oncology of Breast Cancer, Peking University Cancer Hospital & Institute
Other Study IDs: Y-Gilead2024-ZD-0212
Record Dates: First submitted 2025-05-07; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: TNBC
Keywords: sacituzumab govetican; toripalimab; ADC; triple-negative breast cancer; first-line therapy; immune-checkpoint inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; toripalimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue specimens, peripheral blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sacituzumab govitecan combined with Toripalimab
  Interventions: Drug: Sacituzumab Govitecan (SG)+Toripalimab

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG)+Toripalimab — Sacituzumab govitecan (Trodelvy): 10mg/kg, administered by intravenous infusion on day 1 and day 8.
  Toripalimab: 240mg, administered by intravenous infusion on day 1.
  Other Names: IMMU-132; Trodelvy™; GS-0132; Toripalimab

SUMMARY:
The goal of this study is to explore the efficacy and safety of sacituzumab govitecan in combination with toripalimab as first - line treatment in patients with advanced triple - negative breast cancer.

The main questions it aims to answer are:

1. To investigate the efficacy and safety of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer.
2. To explore the biomarkers that can predict the efficacy of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer.

Participants will:

Have their progression - free survival (PFS) observed and evaluated. Have all adverse events and immune - related adverse events monitored to assess safety.

Have their objective response rate measured as a secondary outcome. Have their survival period tracked as a secondary outcome. Have biomarkers associated with efficacy observed and explored as a secondary outcome.

DETAILED DESCRIPTION:
1. Research Objectives： The overall objective of this study is to explore the efficacy and safety of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer.

Primary Objectives：1）To observe and evaluate the efficacy (progression - free survival, PFS) of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer under real - world conditions.2）To observe and evaluate the safety (all adverse events and immune - related adverse events) of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer under real - world conditions. Secondary Objectives：Objective response rate.Survival.To observe and explore biomarkers associated with efficacy. 2. Significance of the Research：Currently, chemotherapy remains the main treatment for advanced triple - negative breast cancer. However, whether it is single - agent or combination chemotherapy, the efficacy is rather poor. Improving the efficacy and safety of first - line treatment for advanced triple - negative breast cancer is an urgent problem to be solved. Both sacituzumab govitecan and toripalimab are major drugs for the treatment of advanced triple - negative breast cancer, and combination therapy may further enhance the effectiveness of treatment. At present, there is no literature reporting the efficacy and safety data of sacituzumab govitecan in combination with toripalimab as first - line treatment. This study is a prospective, single - arm, multicenter, non - interventional, observational clinical trial, aiming to observe the efficacy and safety of sacituzumab govitecan in combination with toripalimab as first - line treatment for advanced triple - negative breast cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients aged 18 to 75 years old;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score: 0 to 1;
3. Patients with histologically or cytologically confirmed advanced triple-negative breast cancer;
4. Patients who have not received systemic treatment (including chemotherapy, targeted therapy and immunotherapy) for advanced triple-negative breast cancer;
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 standard, having at least one measurable lesion;
6. Deciding to receive anti-tumor treatment with the combination of sacituzumab govitecan and toripalimab.

Exclusion Criteria:

1. Patients with symptomatic brain metastases (such as increased intracranial pressure, epilepsy, etc.) who require emergency radiotherapy or surgical intervention;
2. Patients who have previously received HER2-targeted therapy or Trop-2-targeted therapy;
3. Patients who have previously used or are currently using PD-(L)1 inhibitors and/or ADC drugs containing topoisomerase inhibitors, such as sacituzumab govitecan, Dato-DXd, etc., as well as topoisomerase inhibitors;
4. Patients who are considered by the investigator to be unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving first-line treatment for advanced triple-negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Enrollment up for approximately 36 months.
  PFS is defined as the time from the date of randomization until the date of objective progressive disease (PD) or death (whichever comes first).

SECONDARY OUTCOMES:
Overall Survival (OS) | Enrollment up for approximately 53 months.
  OS is defined as the time from the date of randomization until death due to any cause.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | First dose date up to 30 days post last dose, up to approximately 53 months
Objective Response Rate (ORR) as Assessed by BICR per RECIST Version 1.1 | Enrollment up for approximately 53 months.
  ORR is defined as the proportion of participants who achieve complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Percentage of Participants Experiencing Clinically Significant Laboratory and/or Vital Sign Abnormalities | First dose date up to 30 days post last dose, up to approximately 53 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided